CLINICAL TRIAL: NCT03732287
Title: A Phase I Dose Ranging Study Evaluating the Safety and Efficacy of Cooling Anesthesia for Local Anesthesia During Intravitreal Injection (COOL 1)
Brief Title: Cooling Anesthesia for Intravitreal Injection
Acronym: COOL-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Recens Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COOL-1.0
Record Dates: First submitted 2018-11-01; First posted 2018-11-06 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia, Local; Intravitreal Injection; Macular Degeneration; Diabetic Macular Edema
Keywords: intravitreal injection; anesthesia; macular degeneration; diabetic macular edema
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: A dose escalation strategy of differing temperatures and duration to test safety and efficacy of cooling anesthesia for intravitreal injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- -5 degrees Celsius for 10 seconds (Experimental)
  Interventions: Device: Cooling Anesthesia
- -5 degrees Celsius for 20 seconds (Experimental)
  Interventions: Device: Cooling Anesthesia
- -10 degrees Celsius for 10 seconds (Experimental)
  Interventions: Device: Cooling Anesthesia
- -10 degrees Celsius for 20 seconds (Experimental)
  Interventions: Device: Cooling Anesthesia

INTERVENTIONS:
Device: Cooling Anesthesia — Application of cooling anesthesia device prior to intravitreal injection

SUMMARY:
The purpose of this clinical study is to evaluate the safety and efficacy of cooling anesthesia application to the eye as anesthesia for intravitreal injection using a novel cooling anesthesia device and determine the effects of temperature and duration of application on subjective pain after intravitreal injection.

DETAILED DESCRIPTION:
Intravitreal injections have become the standard of care for administering medications for retinal diseases such as age related macular degeneration and diabetic macular edema. There is considerable apprehension among patients receiving these injections, primarily revolving around adequate anesthesia during the injection. Current methods of anesthesia involve topical anesthetic drops, lidocaine gels, or subconjunctival injections of lidocaine, which suffer from either poor anesthetic effect, corneal irritation, or subconjunctival hemorrhage, as well as significant time for the onset of anesthesia.

Recens Medical has developed a novel medical device which can precisely and rapidly cool the surface of the eye This device cools to a temperature around -5 to -10 degrees Celsius, about the temperature of a cold ice cube, and thus has an excellent safety profile compared to conventional ophthalmic cryotherapy units. The value of such a device is both improved patient comfort, as well as increased efficiency and workflow for retina specialists administering intravitreal injections.

This device has been extensively tested in animal safety studies as well as pilot human studies and has not demonstrated any serious adverse effects and has shown anesthetic effects comparable to current standard of care.

This dose escalation study will test various temperatures and duration of temperatures to evaluate for safety as well as determine the optimal temperature for anesthesia during intravitreal injection.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years old at screening visit.
* Men and women who are undergoing intravitreal injections in either one eye or both eyes with either Lucentis or Eylea as part of their normal standard of care with a 30 gauge needle.
* Subject has received a minimum of 3 intravitreal injections in the study eye prior to the study visit.
* Subject is willing and able to sign the study written informed consent form (ICF).

Exclusion Criteria:

* History of presence of scleromalacia
* Preexisting conjunctival, episcleral or scleral defects
* Less than 18 years of age
* Unable to provide informed consent
* Has received less than 3 injections in the study eye
* Active severe eye disease not controlled with artificial tears and requiring Restasis or Xiidra drops.
* History of Endophthalmitis with intravitreal injection
* History of uveitis
* History of retinal detachment in either eye
* History of vitrectomy

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Subjective Pain | 24-48 hours after injection
  Pain as measured by the visual analogue scale (VAS). This was used in the previously presented SOLAR study (Clinical trials.gov, NCT01926977). Total range is 0-10, with 0 being no pain, and 10 being unbearable pain.
Number of patients with treatment adverse events as measured by slit lamp examination | 30 minutes after injection
  Full slit lamp examination of anterior and posterior segment after intravitreal injection

SECONDARY OUTCOMES:
Subject response to needle penetration | Intraoperative (During injection)
  subject response to needle penetration as evaluated by physician
Time to perform intravitreal injection | Intraoperative (injection procedure)
  Time to perform injection, measured from beginning of anesthesia to intravitreal injection

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Khanani, MD, Principal Investigator — Sierra Eye Associates
Locations (2):
- United States (2):
  - Sierra Eye Associates, Reno, Nevada
  - Retina Consultants of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Results of this study will be presented at a national meeting